CLINICAL TRIAL: NCT04462705
Title: Abdominal Massage to Prevent Postoperative Ileus as Part of an Enhanced Recovery Program After Colorectal Surgery
Brief Title: Abdominal Massage to Prevent Postoperative Ileus After Colorectal Surgery
Acronym: MATRAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 38RC20.021
Record Dates: First submitted 2020-02-20; First posted 2020-07-08 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Colorectal Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual physiotherapeutic intervention (Active Comparator): the usual physiotherapeutic intervention (respiratory and walking exercices). Each patients will be treated following the ERAS Guideline.
  - At D + 1 post-surgical:
  1. - First lift with verticalization.
  2. - A session with the Cliniflo® in a seated position.
  3. - Walk at least 100 m with the help of the physiotherapist.
  At- D+2 and D+3 post-surgical Same session as on D+1 with progressive increase in the walking perimeter. Add up and down stairs on D+ 3
  Interventions: Procedure: Usual physiotherapeutic intervention and Abdominal Massage
- abdominal massage and usual physiotherapeutic intervention (Experimental): the usual physiotherapeutic intervention (respiratory and walking exercices). Each patients will be treated following the ERAS Guideline.
  - At D + 1post-surgical:
  1. - First lift with verticalization.
  2. - A session with the Cliniflo® in a seated position.
  3. - Walk at least 100 m with the help of the physiotherapist.
  At- D + 2 and D + 3 post-surgical Same session as on D + 1 with progressive increase in the walking perimeter. Add up and down stairs on D+ 3
  In this experimental arm, a abdominal massage will be performed in addition to the usual physiotherapeutic intervention (respiratory and walking exercices).
  The sessions take place on D+1, D+2 and D+3 post-surgical The first session is performed at least 20 hours after surgery (incision begins) Never within an hour of a meal. The session is timed.
  Interventions: Procedure: Usual physiotherapeutic intervention and Abdominal Massage

INTERVENTIONS:
Procedure: Usual physiotherapeutic intervention and Abdominal Massage — Abdominal massage is not widely applied amongst general surgery team and is not part of the recommendation. This technique refers to profound manœuvrers of visceras through abdominal palpation and breathing, and has been used as part of the local protocol of Grenoble Alps University Hospital for many years with satisfactory results. No complications have been reported.

SUMMARY:
Post operative ileus refers to an disrupt in normal gastrointestinal motility responsible of nausea and vomiting. It occurs in about 15-20% of colorectal surgeries. Some preventive measures have been included in the Enhanced Recovery After Surgery Program such as early mobilisation and enteral feeding or minimal invasive approach.

Abdominal massage is not widely applied amongst general surgery team and is not part of the recommendation. This technique refers to profound manœuvrers of visceras through abdominal palpation and breathing, and has been used as part of the local protocol of Grenoble Alps University Hospital for many years with satisfactory results. No complications have been reported.

Various studies have evaluated the value of physiotherapy and massage for resumption of normal bowel function. A study from Rouen University Hospital demonstrated that a mechanical stress to the cuteaneous tissue by LPG Cellu M50® machine would reduce pain and lower the time to first flatus. Similar results were obtained after Cardiac surgery. In a preclinical study on operated rats, abdominal massage also improved normal bowel function recovery.

Physiotherapist plays a key role in RAC. Their action on respiratory function (movement of diaphragm) and musculoskeletal system (early walking) allows a faster recovery and a reduction of time of hospitalization. Even though the results on time to first flatus and anxiety seem interesting, Deep abdominal massage has never been evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >18years (homme et femme de plus de 18 ans)
* Elective Patients undergoing colorectal surgery with intestinal anastomosis (Colectomy, Anterior Resection, intestinal resection or stoma closure) without protective stoma creation in an Enhanced Recovery After Surgery Program
* Able to give the consent
* Affiliated to Social Security

Exclusion Criteria:

* Mental disorders
* Cutaneous infection on the abdomen
* Pregrancy and breast feeding
* Patients unable to give their free consent (incarcerated, legal protection measures)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2021-09-09 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of abdominal massage on time to normal bowel function after colorectal surgery | through study completion, 30 days
  Time to normal bowel function

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand TRILLING, MD, PhD, Principal Investigator — BTrilling@chu-grenoble.fr
Locations (1):
- CHu grenoble alpes, Grenoble, France

REFERENCES:
- [Background] Le Blanc-Louvry I, Costaglioli B, Boulon C, Leroi AM, Ducrotte P. Does mechanical massage of the abdominal wall after colectomy reduce postoperative pain and shorten the duration of ileus? Results of a randomized study. J Gastrointest Surg. 2002 Jan-Feb;6(1):43-9. doi: 10.1016/s1091-255x(01)00009-9. PMID 11986017
- [Background] Bauer BA, Cutshall SM, Wentworth LJ, Engen D, Messner PK, Wood CM, Brekke KM, Kelly RF, Sundt TM 3rd. Effect of massage therapy on pain, anxiety, and tension after cardiac surgery: a randomized study. Complement Ther Clin Pract. 2010 May;16(2):70-5. doi: 10.1016/j.ctcp.2009.06.012. Epub 2009 Jul 14. PMID 20347836
- [Background] Dreyer NE, Cutshall SM, Huebner M, Foss DM, Lovely JK, Bauer BA, Cima RR. Effect of massage therapy on pain, anxiety, relaxation, and tension after colorectal surgery: A randomized study. Complement Ther Clin Pract. 2015 Aug;21(3):154-9. doi: 10.1016/j.ctcp.2015.06.004. Epub 2015 Jun 12. PMID 26256133
- [Background] Chapelle SL, Bove GM. Visceral massage reduces postoperative ileus in a rat model. J Bodyw Mov Ther. 2013 Jan;17(1):83-8. doi: 10.1016/j.jbmt.2012.05.004. Epub 2012 Aug 12. PMID 23294688
- [Background] Navalgund A, Axelrod S, Axelrod L, Singhal S, Tran K, Legha P, Triadafilopoulos G. Colon Myoelectric Activity Measured After Open Abdominal Surgery with a Noninvasive Wireless Patch System Predicts Time to First Flatus. J Gastrointest Surg. 2019 May;23(5):982-989. doi: 10.1007/s11605-018-4030-4. Epub 2018 Nov 2. PMID 30390183